CLINICAL TRIAL: NCT00831038
Title: A Pilot Study of Pulmonary Function in Dysphagic Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, James D. Tutor, M.D., James D. Tutor, M.D., University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#8819
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Lung Disease
Keywords: pulmonary function tests; infants; chronic lung disease; dysphagia; chronic aspiration
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Infant Pulmonary Function Tests — Tests will be performed on study patients within 1 week of study enrollment and again 6 months later.

SUMMARY:
Infants less than 2 years old who have been newly diagnosed with problems swallowing will have pulmonary function tests performed to try to detect the presence of chronic lung disease. Six months later after the infants have received appropriate therapy for their swallowing problems, pulmonary function tests will be performed again to see if there has been any change in their chronic lung disease.

DETAILED DESCRIPTION:
Twenty-five infants between the ages of 1 month and 24 months who have just been diagnosed with dysphagia via a modified barium feeding study will be recruited into the study. The infants will be sedated with chloral hydrate and have pulmonary functions measured (pre- and post-bronchodilator spirometry and lung volume) using the infant pulmonary laboratory. Treatment for the infants' dysphagia/chronic aspiration will be treated as determined by the primary care physicians. Six months later the infants will again be sedated and have pulmonary functions measured. Results of the two sets of tests will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* infants between ages 1-24 months who have been newly diagnosed with dysphagia

Exclusion Criteria:

* cystic fibrosis
* obstructive sleep apnea
* seizures
* allergy or adverse reaction to chloral hydrate
* heart disease
* liver disease
* kidney disease
* pneumonia
* pleural effusion
* neuromuscular disease
* major congenital anomalies
* tracheoesophageal fistula
* vascular ring
* bronchopulmonary dysplasia
* pharyngeal anomalies
* Arnold-Chiari malformation

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
infant pulmonary function test results | On admission to study and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: James D Tutor, MD, Principal Investigator — Methodist/LeBonheur Healthcare/University of Tennessee College of Medicine
Locations (1):
- LeBonheur Children's Medical Center, Memphis, Tennessee, United States